CLINICAL TRIAL: NCT05023642
Title: Training-induced Muscle Strength Increase and Its Role in Interface Pressure in Inelastic Compression: A Randomized Clinical Trial
Brief Title: Training-induced Muscle Strength and Its Role in Interface Pressure in Inelastic Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pró Circulação® (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Strengthinelastic
Record Dates: First submitted 2021-08-09; First posted 2021-08-26 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Resistance Training
Keywords: Inelastic compression; Resistance exercise; Muscle hypertrophy; Chronic venous disease
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers who will perform both pre and post-test evaluations, as well as data analysis, will be blinded regarding randomization. Blinding will be ensured by asking investigators at the end of the trial if investigators knew the arm to which each subject will be allocated prior to opening the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- resistance training (Experimental): Participants will not be offered the exercise program in the three months before data collection.
  From then on, participants will perform exercises during the resistance training protocol intervention.
  Interventions: Other: resistance training
- control group (No Intervention): Individuals in the control group will not be offered the exercise program in the three months before data collection and during the entire period corresponding to the 12-week intervention.

INTERVENTIONS:
Other: resistance training — Interventions will include a three-phase strengthening training protocol.
  1. Adaptation phase: three sessions, emphasis on learning the technique, body self-awareness, and movement coordination;
  2. Basic phase: 12 sessions, to increase muscle strength; and
  3. Specific phase: 21 sessions, to intensify the process of strength gain and muscular hypertrophy.
  Participants will perform the following exercises during the strength-training protocol intervention: pec deck/seated lever fly, adductor, pulldown, abductor strengthening, alternating dumbbell curl, leg press at a 45-angle, triceps pulley, lateral raise, knee flexion and extension, ankle joint flexion and extension in the leg press, and crunches. If the participant has difficulty performing a specific exercise, an equivalent activity will replace it. From the eighth week onwards, participants will perform additional exercises focused on strengthening the gastrocnemius and soleus.
  Arms: resistance training

SUMMARY:
The present study will answer the following question: what are the effects of strength gain and muscle hypertrophy on interface pressure, static stiffness index, and working pressure amplitude in the elderly using inelastic compression?

DETAILED DESCRIPTION:
This phase I two-armed randomized clinical trial including participants above 60 years of age who do not present any musculoskeletal limitations preventing their participation in resistance exercise programs will be conducted at the Ativas Gym, Xanxere/SC, Brazil. Participants will perform exercises during the strength-training protocol intervention, while individuals in the control group will not be offered the exercise program in the three months before data collection and during the entire period corresponding to the 12-week intervention. In addition, we will monitor their eating and physical activity habits throughout the data collection period. The study was designed in accordance with the CONSORT statement.

ELIGIBILITY:
Inclusion Criteria:

* Participants above 60 years of age who do not present any musculoskeletal limitations preventing their participation in strengthening exercise programs.

Exclusion Criteria:

* Participants who present chronic venous insufficiency (CEAP C3-6) evaluated through Doppler ultrasonography, severe congestive heart failure (functional class III and IV - NYHA), and Ankle/Brachial Index (ABI) < 0.8. We will also exclude elderly individuals who are unable to perform the required exercises due to physical limitations and those bedridden or wheelchair-bound.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline body composition at 12 weeks | Baseline visit and follow-up after 12 weeks
  The body composition assessment will be performed through Dual-Energy X-Ray Absorptiometry (DXA) examination, on the first and last day of the study, in both groups, with the participant fasting, without having exercised in the last 24 hours (Andreoli et., 2009).
Change from baseline muscle strength at 12 weeks | Baseline visit and follow-up after 12 weeks
  Muscle strength assessments will be performed at the beginning and end of the intervention (pre-test and post-test) in all study participants. After warming up the lower limbs, based on dynamic movements, for three minutes, each participant will perform between six and eight repetitions with 50% of the estimated maximum load and, one minute later, three repetitions with 70% of the estimated load. Three minutes after the specific warm-up, the test will start. An interval of two minutes will be considered between each attempt, and no more than five attempts will be made for each participant. The load corresponding to the last successful attempt will be considered as a result (Brown & Weir, 2001).
Change from baseline handgrip strength at 12 weeks | Baseline visit and follow-up after 12 weeks
  We will perform the handgrip test assessments at the beginning and end of the intervention (pre-test and post-test) in all study participants. We will use a dynamometer in the sitting position, with the shoulder slightly adducted, elbow flexed to 90º, forearm in a neutral position, and, finally, the position of the wrist can vary from 0 to 30º of extension. Three 3-second isometric muscle contractions will be performed, in order to record the handgrip strength obtained (Fernandes & Marins, 2011).
Change from baseline walking speed at 12 weeks | Baseline visit and follow-up after 12 weeks
  We will perform walking speed assessments at the beginning and end of the intervention (pre-test and post-test) in all study participants. Will be evaluated through the test of walking speed of 4 meters, participants will perform the test walking with normal stride speed throughout the course (Braden, 2012).
Change from baseline interface pressure at 12 weeks | Baseline visit and follow-up after 12 weeks
  We will measure the interface pressure exerted by the bandage/velcro device at point B1 (the area located at the transition between the Achilles tendon and the muscular portion of the medial gastrocnemius muscle). We will perform the interface pressure assessments at the beginning and end of the intervention (pre-test and post-test) in all study participants using a PicoPress pneumatic system.
Change from baseline Static Stiffness Index at 12 weeks | Baseline visit and follow-up after 12 weeks
  Static Stiffness Index will be calculated by the difference in the interface pressure measure between the supine and standing positions, at the beginning and end of the intervention (pre-test and post-test).
Change from baseline Working Pressure Amplitude at 12 weeks | Baseline visit and follow-up after 12 weeks
  Working Pressure Amplitude (WPA) will be considered as the difference between the lowest and highest interface pressure recorded during flexion and extension movements of the ankle joint and during walking. And will be performed at the beginning and end of the intervention (pre-test and post-test).

SECONDARY OUTCOMES:
Change from quality of life assessment at 12 weeks | Baseline visit and follow-up after 12 weeks
  The Short-Form 36 (SF-36) questionnaire will be used; scores will be assigned to each question. Changing the scale from zero to 100, values closer to zero being considered a negative perception of quality of life and close to 100 as a positive perception of quality of life (Ciconelli et al., 1999).
Change from baseline lower limbs' functional strength at 12 weeks | Baseline visit and follow-up after 12 weeks
  We will evaluate lower limbs' functional strength at the beginning and end of the intervention (pre-test and post-test) in all study participants. Using the Chair-test, it will be measured using a chair without armrests with a seat height of approximately 43 cm from the floor. The test will start with the participant sitting in the middle of the chair. At the signal, the participant will rise to full extension of the knee joint (upright body) and then return to the starting sitting position (Jones et al., 1999).
Change from baseline dynamic balance at 12 weeks | Baseline visit and follow-up after 12 weeks
  It will be performed using the timed up and go test. The test consists of getting up from a chair, going around a cone three meters away, and sitting back down on the chair. The time it takes the subject to get up from a chair, walk, return to the chair and sit down again is recorded (Podsiadlo & Richardson, 1991).

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Matta, MD, Principal Investigator — Pró Circulação®; Clodoaldo A. De Sá, Ph.D., Principal Investigator — Unochapecó
Locations (2):
- Brazil (2):
  - Unochapecó University, Chapecó, Santa Catarina
  - Pró Circulação® - Clinic of Angiology and Vascular Surgery, Xanxerê, Santa Catarina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreoli A, Scalzo G, Masala S, Tarantino U, Guglielmi G. Body composition assessment by dual-energy X-ray absorptiometry (DXA). Radiol Med. 2009 Mar;114(2):286-300. doi: 10.1007/s11547-009-0369-7. Epub 2009 Mar 5. English, Italian. PMID 19266259
- [Background] Brown LE, Weir JP. Asep procedures recommendation I: accurate assessment of muscular strength and power. Journal of Exercise Physiology Online. 2001;4:1-21.
- [Background] Fernandes, A.A., Marins, J.C.B.. Teste de força de preensão manual: analise metodológica e dados normativos em atletas. Fisoter Mov. 2011;24(3):567-78.
- [Background] Braden, H. Self-selected gait speed: A critical clinical outcome. Lower Extremity Review. 2012 Nov.
- [Background] Ciconelli, RM, et al. Tradução para a língua portuguesa e validação do questionário genérico de avaliação de qualidade de vida SF-36 (Brasil SF-36). Ver Bras Reumatol. 1999;39(3):143-150.
- [Background] Yim E, Richmond NA, Baquerizo K, Van Driessche F, Slade HB, Pieper B, Kirsner RS. The effect of ankle range of motion on venous ulcer healing rates. Wound Repair Regen. 2014 Jul-Aug;22(4):492-6. doi: 10.1111/wrr.12186. PMID 25041619
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Rubin RW, Maher M. Actin turnover during encystation in Acanthamoeba. Exp Cell Res. 1976 Nov;103(1):159-68. doi: 10.1016/0014-4827(76)90251-2. No abstract available. PMID 991946
- [Background] Da Matta, E.S. et al. A Combined Therapy Protocol to Improve Lower Extremity Muscle Pumping Function and Lymphatic Drainage for Venous Ulcer Healing. J Vasc Med Surg. 2017;5:347. Doi: 10.4172/2329-6925.1000347
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946